CLINICAL TRIAL: NCT02119338
Title: Barrow ALA Trial for Recurrent Gliomas
Brief Title: 5-ALA in Recurrent Glioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11BN092
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Glioma
Keywords: 5-ala; 5-aminolevulinic acid; fluorescence-guided surgery; glioma; astrocytoma; glioblastoma; oligodendroglioma; recurrence of glioma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma; Oligodendroglioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-ala preoperatively (Experimental): A dose of 5-ala will be taken by mouth approximately 3 hours before going to surgery.
  Interventions: Drug: 5-ala

INTERVENTIONS:
Drug: 5-ala — dose of 5-ala will be taken as either 5 mg/kg, 10 mg/kg, or 20 mg/kg approximately 3 hours before going to surgery.
  Other Names: 5-aminolevulinic acid; Levulin(R)

SUMMARY:
The investigators propose a single-center, non-randomized, single-arm study at the Barrow Neurological Institute/St. Joseph's Hospital for recurrent glioma. The 5-ALA for recurrent glioma study will correlate presence of fluorescence in tumor tissue with pathological findings. This will be done using three cohorts in dose escalation. The investigators' hypothesis is that (for both low- and high-grade gliomas,) a lower dose of 5-ALA will result in less false positive fluorescence.

DETAILED DESCRIPTION:
The goal is to determine the dose of 5-ALA which promotes the lowest volume of residual disease after resection of recurrent high grade glioma without compromising the demarcation between recurrent high grade glioma and postoperative bed normal tissue.

Sub-goals:

1. To determine the impact of the dose of 5-ALA in improving volumetric extent of resection in patients with recurrent high grade gliomas
2. To determine the impact of the dose of 5-ALA in improving overall survival of recurrent high grade glioma patients
3. To determine the impact of the dose of 5-ALA in improving progression-free survival of recurrent high grade glioma patients
4. To determine the impact of the dose of 5-ALA on the neurological morbidity of recurrent high grade glioma patients.

Patients with presumed recurrent glioma will be entered into the trial. Those with recurrent disease will receive study drug (5-ALA) in one of three dose-escalated cohorts (5 mg/kg; 10 mg/kg; 20 mg/kg). Intraoperatively, patients will undergo resection with combined fluorescence microscopy and confocal microscopy. Resected tissue specimens corresponding to the presence of fluorescence will be sent to pathology for examination. Postoperatively, patients will have an MRI with and without contrast within 48 hours of surgery. Subsequent analysis of each patient will include assessment of the primary endpoint (volume of residual disease) by volumetrically quantifying the tumor before and after surgery using T1-weighted contrast-enhancement. Similarly, volumetric extent of resection will also be measured.

ELIGIBILITY:
Inclusion Criteria

* Presumed recurrent glioma
* Age > 18 years
* Normal bone marrow function (WBC > 3000, Platelets > 100,000)

Exclusion Criteria

* Pregnancy
* History of photosensitivity, porphyria, or exfoliative dermatitis
* Hepatic dysfunction in the last 12 months [defined by aspartate aminotransferase(AST), alanine aminotransferase (ALT) , alkaline phosphatase (ALP) , bilirubin > 2.5 x normal]
* Serum creatinine > 180 µmol/L
* Estimated Glomerular Filtration Rate (eGFR)< 60 ml/min/1.73m2
* Inability to undergo MRI with contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Presence of fluorescence in tumor tissue compared to tissue with treatment effect. | day of surgery-1 day
  Correlation of fluorescence with pathological findings

SECONDARY OUTCOMES:
Extent of resection | time within 48 hours post operative
  A postoperative MRI with contrast will be acquired within 48 hours of surgery. Volumetric analysis of contract T1-weighted images (for low grade gliomas) will be compared to the preoperative sequences to calculate the volume of residual disease. Slice-by-slice assessment of pre- and postoperative tumor volume will be quantified by sequentially measuring the area of tumor on each slice and then integrating the combined measurements. This methodology has been previously reported (Sanai et al., Journal of Neurosurgery, 2010; Sanai et al, The New England Journal of Medicine, 2008)
Progression-free survival rate at 6 months | time from date of surgery to 6 months post surgery
Overall survival | time from date of surgery to date of death from any cause, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Barrow Neurosurgical Associates
Locations (1):
- Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States